CLINICAL TRIAL: NCT06549270
Title: Unraveling the Spectrum of Migraine Resistant to Treatments: Searching for Novel Biological PHEnotypes and theRApeutic Approaches (SPHERA Project)
Brief Title: Biochemical Profiling of Migraine Patients
Acronym: SPHERA_WP1_1
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of L'Aquila (Other)
Responsible Party: Sponsor
Other Study IDs: SPHERA- eCBome
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Migraine Disorders; Chronic Migraine; Episodic Migraine
Keywords: migraine; anti CGRP mABs; calcitonin gene related peptide; endocannabinoid system
MeSH Terms: conditions — Migraine Disorders | interventions — Ligands

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: Patients with high frequency episodic migraine (HFEM) or chronic migraine (CM) undergoing treatment with monoclonal antibodies directed against calcitonin gene related peptide pathway (mAbs) who obtained a reduction in monthly migraine days equal or higher than 50% after three months of treatment compared to pre-treatment values.
  Interventions: Drug: MAbs
- Non-Responders: Patients with HFEM or CM undergoing mAbs treatment who obtained a reduction in monthly migraine days < 50% after three months of treatment compared to pre-treatment values.
  Interventions: Drug: MAbs

INTERVENTIONS:
Drug: MAbs — Monthly or quarterly mAbs administration
  Other Names: Monoclonal antibody targeting the CGRP pathway (ligand or receptor) (mAbs)

SUMMARY:
Aim of the study was to assess a potential dysfunction of the endocannabidiome system (eCBome) in migraine patients. Migraine patients who will undergo preventive therapy with monoclonal antibodies directed against the calcitonin gene related peptide (mAbs) will be evaluated through a deep phenotyping of peripheral neurochemical biomarkers (eCBome, neuropeptides, cytokines and kynurenine levels, and microRNAs expression).

Primary aim is to assess baseline differences among those patients who achieved a reduction of monthly migraine days >/= 50% after three months of tretament (namely Responders) and those who did not (namely Non-responders).

DETAILED DESCRIPTION:
Previous evidence showed that endocannabidiome system (eCBome) is altered in migraine patients demonstrating: i) altered gene expression of catabolizing enzymes (MAGL and FAAH) in patients with episodic and chronic migraine compared to healthy controls; ii) altered peripheral levels of the endocannabinoid-like lipid palmitoylethanolamide (PEA) with evidence of increased PEA levels during the acute migraine phase.

Despite the high effectiveness and tolerability of mAbs monoclonal antibodies directed against the Calcitonin gene related peptide (mAbs), evidence from RCTs and real-life studies demonstrates that mAbs fail in 40% of patients. These patients may bear a non CGRP- dependent phenotype, potentially linked to eCBome dysfunction.

Primary aim is to perform a deep phenotyping of the whole cohort of migraine patients comparing the subgroups of those patients who will be Responders to mAbs treatment (namely those patients who achieved a reduction of monthly migraine days >/= 50%) compared to the Non-Respoder group (namely those patients who achieved a reduction of monthly migraine days < 50%) .

Neuropeptides, microRNAs, inflammatory cytokines, and kynurenine metabolites will be evaluated. These findings will allow the identification of a multibiomarkers panel signature of migraine patients resisting to specifically targeted preventive treatments and potentially unveiling other molecular targets.

STUDY DESIGN:

This study is part of the SPHERA project with funding from the Italian Ministry of Health (GR-2021-12372429). Patients will be enrolled from those attending the outpatient clinic of IRCCS Mondino Institute (Pavia) and Neurology Department of the University of L'Aquila (Avezzano).

Data will be collected before mAbs starting (baseline-T0) and after three months (T1) of mAbs treatment. First, Repsonder and Non-responder groups will be identified, then a biochemical profiling of the two subgroups will be performed at T0 and T1.

METHODS:

All patients will undergo a biochemical profiling that will include analysis of:

* eCBome system: mRNS levels of FAAH, MAGL, DAGL, NAPE, NAAA in peripheral blood mononuclear cells,
* plasma levels of AEA, 2-AG, PEA and OEA; CGRP, PACAP, and VIP; IL-1beta, TNF-alpha, IL-4, and IL-10; kynurenic and quinolinic acids;
* miR-382-5p, miR-34a, miR-30a, and miR-155 in peripheral blood mononuclear cells,
* shotgun analysis of microbiota in patients' faeces.

Biochemical sampling will be collected between 9 and 11 a.m. to avoid circadian rhythm influence. All evaluation will be performed in migraine interictal phase.

The following collection methods will be adopted:

* mRNA and microRNA analysis in PBMCs. Blood samples will be collected within ethylenediamine tetra-acetic acid tubes, with a first isolation of PBMCs and total RNA. Ubiquitin C and U6 will act as housekeeping genes for genes coding for the eCBome enzymes and miRNAs.
* kynurenic acid and quinolinic acid, AEA, PEA, 2-AG and OEA will be determined according to Gao published method (Gao, 2020). Kinurenine metabolite levels will be measured according to the method described by Fuertig (Fuertig, 2016).
* CGRP alpha, PACAP-38 and VIP levels will be measured using a commercial enzyme linked immunosorbent assay
* IL-1beta, TNF-alpha, IL-4, IL-10 cytokine will be measured by the Ella Automated Immunoassay System with a Simple Plex assay panel.
* Microbiome analysis: after correct collection and preservation of stool specimens, they will be delivered to the Translational Neurovascular Research Unit (IRCCS Mondino Foundation) for DNA extraction.

STATISTICAL ANALYSIS Sample size calculation is defined for primary outcome (MAGL expression), while a power analysis is performed for the co-primary outcome (FAAH expression).

According to preliminary data from the work of Greco 2021 suggesting a ratio between Non-responders and Responders: 2:3 and MAGL gene expression: 8±10 RQ in Non-responders and 3±4 RQ in Responders, the minimum sample size is of 88 migraine patients (53 Responders and 35 NON-Responders) in order to have a confidence interval 95% and power of 80%.

Normality analysis will be performed to evaluate parametric or non-parametric methods.

A univariate analysis will be performed to search for differences in demographic, clinical and biochemical parameters between Non-Responder and Responder groups at T0. Main statistical analysis will include a multivariate approach to control for confounders. The level of significance will be set at alpha = 0.05 considering correction for multiple comparisons where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients aged 18 to 75 years
* diagnosis of episodic migraine or chronic migraine according to ICHD-3 criteria
* for episodic migraine: 8-14 monthly migraine days in the previous 3 months
* diagnosis of resistant migraine defined by: i) having failed at least 3 classes of migraine preventatives and ii) suffering from at least 8 debilitating monthly headache days for at least 3 consecutive months
* patients naive to CGRP targeting treatments

Exclusion Criteria:

* history of major psychiatric or other neurological conditions
* diagnosis of other primary or secondary headache disorders (only sporadic tension-type headache is allowed if the patients can clearly differentiate between the 2 types of headaches)
* changes in ongoing preventive treatment (if any) in the previous 3 months
* clinically significant medical conditions
* chronic pain conditions
* alcohol and/or drug abuse
* pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic or high frequency episodic migraine attending the outpatient clinic of the Headache Science & Neurorehabilitation Unit of the IRCCS Mondino Foundation (Pavia, Italy) and the Neurology Department of the University of L'Aquila (Avezzano, Italy).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Gene expression of FAAH | Baseline (T0) - three months of mAbs treatment (T1)
  Baseline differences in gene expression of fatty acid amide hydrolase (FAAH) in peripheral blood mononuclear cells (PBMC) (continuous variable)
Gene expression of MAGL | Baseline (T0) - three months of mAbs treatment (T1)
  Gene expression of Monoacylglycerol lipase (MAGL) in peripheral blood mononuclear cells (PBMC) (continuous variable)

SECONDARY OUTCOMES:
Gene expression of catalyzing enzymes (DAGL, NAPE, NAAA) | Baseline (T0) - three months of mAbs treatment (T1)
  Gene expression of diacylglycerol lipase (DAGL), N-acylphosphatidyl ethanolamide (NAPE) and N-acylethanolamine acid amidohydrolase (NAAA) in peripheral blood mononuclear cells (PBMC) (continuous variable)
Plasma levels of AEA, 2-AG, PEA, OEA | Baseline (T0) - three months of mAbs treatment (T1)
  Plasma levels of endocannabinoids and related lipids (N-arachidonoyl ethanolamide (AEA), 2-arachidonoyl glycerol (2-AG), PEA and anorexigenic oleoyl ethanolamide (OEA (continuous variable)
Plasma levels of CGRP, PACAP and VIP | Baseline (T0) - three months of mAbs treatment (T1)
  Plasma levels of neuropeptides: calcitonin gene related pepetide (CGRP), pituitary adenylate cyclase-activating peptide (PACAP), vasoactive intestinal peptide (VIP) (continuous variable)
Gene expression of miR-382-5p, miR-34a, miR-30a and miR-155 | Baseline (T0) - three months of mAbs treatment (T1)
  microRNAs gene expression (specifically miR-382-5p, miR-34a, miR-30a and miR-155) in peripheral blood mononuclear cells (PBMC) (continuous variable)
Plasma levels of IL-1beta, TNF-alpha, IL-4 and IL-10 | Baseline (T0) - three months of mAbs treatment (T1)
  Plasma levels of proinflammatory (IL-1beta, TNF-alpha) and anti-inflammatory cytokines (IL-4 and IL-10) (continuous variables)
Plasma levels of kynurenic acid and quinolinic acid | Baseline (T0) - three months of mAbs treatment (T1)
  Plasma levels of kynurenine metabolites (continuous variables)
Shotgun analysis of microbiota | Baseline (T0) - three months of mAbs treatment (T1)
  Shotgun analysis of microbiota in patients' faeces

CONTACTS AND LOCATIONS:
Locations (1):
- Headache Science & Neurorehabilitation Unit, Pavia, Italy

REFERENCES:
- [Background] Gao W, Walther A, Wekenborg M, Penz M, Kirschbaum C. Determination of endocannabinoids and N-acylethanolamines in human hair with LC-MS/MS and their relation to symptoms of depression, burnout, and anxiety. Talanta. 2020 Sep 1;217:121006. doi: 10.1016/j.talanta.2020.121006. Epub 2020 Apr 9. PMID 32498885
- [Background] Fuertig R, Ceci A, Camus SM, Bezard E, Luippold AH, Hengerer B. LC-MS/MS-based quantification of kynurenine metabolites, tryptophan, monoamines and neopterin in plasma, cerebrospinal fluid and brain. Bioanalysis. 2016 Sep;8(18):1903-17. doi: 10.4155/bio-2016-0111. Epub 2016 Aug 15. PMID 27524289
- [Background] Greco R, Demartini C, Zanaboni AM, Tumelero E, Icco R, Sances G, Allena M, Tassorelli C. Peripheral changes of endocannabinoid system components in episodic and chronic migraine patients: A pilot study. Cephalalgia. 2021 Feb;41(2):185-196. doi: 10.1177/0333102420949201. Epub 2020 Sep 23. PMID 32967434
- [Background] De Icco R, Greco R, Demartini C, Vergobbi P, Zanaboni A, Tumelero E, Reggiani A, Realini N, Sances G, Grillo V, Allena M, Tassorelli C. Spinal nociceptive sensitization and plasma palmitoylethanolamide levels during experimentally induced migraine attacks. Pain. 2021 Sep 1;162(9):2376-2385. doi: 10.1097/j.pain.0000000000002223. PMID 33587406